CLINICAL TRIAL: NCT06909136
Title: A Phase Ib/II Clinical Study to Evaluate the Safety , Efficacy and Pharmacokinetics of WJ01024 Tablets Combined With Ruxolitinib Tablets in Patients With Myelofibrosis
Brief Title: A Study to Evaluate Safety , Efficacy and Pharmacokinetics of WJ01024 Tablets Combined With Ruxolitinib in Patients With Myelofibrosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS110-003-Ib/II
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Intermediate- and High-risk Myelofibrosis (MF) Patients With Splenomegaly

STUDY DESIGN:
Intervention Model Description: The study consisted of two phases: Phase Ib and Phase II. Phase Ib was dose expansion of WJ01024 tablets combined with Ruxolitinib tablets.
  Phase II was efficacy expansion of WJ01024 tablets combined with Ruxolitinib tablets.
Masking Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WJ01024 tablet (Experimental): If needed, additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: Ruxolitinib phosphate tablet（Jakavi,NOVARTIS,9104733)

INTERVENTIONS:
Drug: Ruxolitinib phosphate tablet（Jakavi,NOVARTIS,9104733) — 5-20mg BID (dosage per investigator judgement,JAKi intolerable pts will receive recuded dose of RUX(≥ 5mg BID),and suboptimal JAKi response pts will receive RUX of 15-20 mg BID）

SUMMARY:
This is a Phase Ib/II clinical study to evaluate the safety , efficacy and pharmacokinetics of WJ01024 tablets combined with Ruxolitinib tablets in patients with myelofibrosis.The study will be conducted in two phases: Phase 1b and Phase 2.Phase Ib is a dose extension study of WJ01024 tablets combined with ruxolitinib tablets. It is planned to recruit patients with medium to high-risk myelofibrosis accompanied by splenomegaly who have had poor response or intolerance to the previously approved JAK inhibitors for myelofibrosis. Phase II is the efficacy extension stage of WJ01024 tablets combined with ruxolitinib Tablets. It is planned to expand two groups of people. Group A will expand to recruit patients with medium-high risk of myelofibrosis accompanied by splenomegaly who have not responded well to the previously approved JAK inhibitors for myelofibrosis. Group B expanded to recruit patients with medium-high-risk myelofibrosis accompanied by splenomegaly who were intolerant after treatment with previously approved JAK inhibitors for myelofibrosis.

DETAILED DESCRIPTION:
Ruxolitinib tablets have been approved in China since April 2017 as the first-line treatment for most intermediate- and high-risk myelofibrosis (MF) patients with splenomegaly. Compared with supportive treatment alone, ruxolitinib tablets have the efficacy of reducing spleen size and improving the symptoms of myelofibrosis, as well as reducing the risk of death and prolonging the survival of MF patients.Although the clinical efficacy of Ruxolitinib tablets has been confirmed, only about half of MF patients can achieve the ideal therapeutic effect (≥35% reduction in spleen volume and ≥50% improvement in disease symptoms at 24 weeks). Therefore, there is an urgent need for innovative drugs that can be combined with Ruxolitinib tablets to enhance therapeutic efficacy and meet clinical needs.

WJ01024 is a small molecule inhibitor of XPO-1, belonging to the same target small molecule compounds as Selinexor. Compared with Selinexor, the metabolism rate of this product is faster, which can reduce the toxicity in the body. In the Ba/F3-EPOR-JAK2-V617F cell model, the combination of this product and ruxolitinib tablets can enhance its anti-cell proliferation activity. In a clinical study initiated by researchers, this product has shown preliminary efficacy as a monotherapy in patients with myelofibrosis who have relapsed, are refractory to, or intolerant of JAK inhibitors, and is expected to have fewer toxic and side effects than drugs targeting the same site. Based on this, the following research is planned.

This is a Phase Ib/II clinical study to evaluate the safety , efficacy and pharmacokinetics of WJ01024 tablets combined with Ruxolitinib tablets in patients with myelofibrosis.The study will be conducted in two phases: Phase 1b and Phase 2.

Phase Ib is a dose extension study of WJ01024 tablets combined with ruxolitinib tablets. It is planned to recruit patients with medium to high-risk myelofibrosis accompanied by splenomegaly who have had poor response or intolerance to the previously approved JAK inhibitors for myelofibrosis.

Phase II is the efficacy extension stage of WJ01024 tablets combined with ruxolitinib Tablets. It is planned to expand two groups of people. Group A will expand to recruit patients with medium-high risk of myelofibrosis accompanied by splenomegaly who have not responded well to the previously approved JAK inhibitors for myelofibrosis. Group B expanded to recruit patients with medium-high-risk myelofibrosis accompanied by splenomegaly who were intolerant after treatment with previously approved JAK inhibitors for myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the study after receiving full informed consent and sign informed consent;
* Age ≥18 years old, gender unlimited;
* Patients diagnosed with primary myelofibrosis (PMF) according to WHO criteria (2016 edition), or with ET secondary myelofibrosis (PET-MF) or PV secondary myelofibrosis (PPV-MF) according to International Working Group on Myelofibrosis Research and Treatment (IWG-MRT) criteria; They could be included regardless of JAK2 mutation；
* Participants with international prognostic scoring system (DIPSS) risk category of intermediate-1, or intermediate-2, or high-risk；
* ECOG score 0~2;
* No stem cell transplantation plan in the near future;
* Spleen enlargement:palpable splenomegaly(≥5cm below left costal margin)or radiologically confirmed spleen volume ≥450 cm^3 using MRI/CT;
* Patients with intolerance or a suboptimal response to prior JAK inhibitor therapy；
* Sufficient hematology and organ function；

Exclusion Criteria:

* More than 10% blasts in peripheral blood or bone marrow；
* Previous treatment with XPO1 inhibitors；
* Unable to cooperate with or unable to perform MRI or CT scans as deemed necessary by sponsor and investigator；
* Treatment with a powerful CYP3A inhibitor or inducer within 14 days prior to initial administration；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
AE | 3 years
  Incidence rate and severity of adverse events and serious adverse events,as well as abnormal changes in clinical significance laboratory tests and other examinations
SVR35 | 3 years
  At weeks 12 and 24, the ratio of splenic volume reduction ≥35% (SVR35) was assessed by the investigator
The absolute value changes of the total symptom score in MPN-SAF-TSS | 3 years
  The absolute value changes of the overall symptom score in MPN-SAF-TSS based on subject assessment in weeks 12 and 24 compared with the baseline

SECONDARY OUTCOMES:
The blood concentration of WJ01024 | 1.5 years
  AUC of WJ01024,C1D1,C2D1,C4D1,C6D1 1 h after WJ01024 administration Both in phase Ib and II
Incidence rate and severity of adverse events nd serious adverse events | 3 years
  Incidence and severity of adverse events nd serious adverse events,as well as abnormal changes in clinical significance laboratory tests and other examinations
Anemia response rate | 3 years
  Anemia response rate at Week 12 and Week 24 as assessed by the investigator according to IWG-MRT criteria
ORR：CR + PR + clinical improvement | 3 years
  Overall response rate (ORR, CR + PR + clinical improvement) as determined by the investigator according to IWG-MRT criteria
PFS | 3 years
  PFS as assessed by the investigator
OS | 3 years
  Overall survival
LDH | 3 years
  Evaluation of changes in serum LDH levels
Phase II：The rate of a reduction of ≥50% in the total symptom score in MPN-SAF-TSS | 3 years
  The rate of a reduction of ≥50% in the overall symptom score in MPN-SAF-TSS based on subject assessment in weeks 12 and 24 compared with the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Zhengzhou, China